CLINICAL TRIAL: NCT03556527
Title: Long-term Radiographic and Clinic Outcomes of Ulnar Shortening Osteotomy in Patients With Ulnar Impaction Syndrome and Reverse Oblique Sigmoid Notch
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-05-005CC
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-04

CONDITIONS: Distal Radioulnar Joint
Keywords: osteotomy; reverse oblique sigmoid notch; ulnar impaction syndrome; ulnar shortening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with ulnar impingement are often coexisting with patients with distal ulnar and ulnar joints with a type of sigmoid notch, and ulnar shortening surgery is one of the most useful and long-lasting treatments for the treatment of ulnar impingement. Some theories point out that if ulnar shortening surgery is performed on patients with distal oblique ulnar incisional ulnar joints, it may lead to accelerated degeneration of distal ulna and ulna articular joints, resulting in worse wrist function. Some theories have pointed out this Instead, surgery will cause joint remodeling and adaptation, but no long-term studies have confirmed this. Therefore, this study plans to evaluate the long-term radiological and clinical outcomes of ulnar shortening surgery performed on patients with preexisting inverted sigmoid notch to determine whether this surgery will cause accelerated distal degeneration of the phalangeal joints or Reshaping of joints and clinically corresponding changes in results.

ELIGIBILITY:
Inclusion Criteria:

* The distal ulnar joint of the wrist contains a patient with an inverted sigmoid notch of the sacrum, and the ulnar impaction causes ulnar wrist pain. Therefore, the ulnar shortening surgery is accepted.

Exclusion Criteria:

* Patients with diagnosed diseases of immune rheumatism, patients with ischemic necrosis of the carpus, patients with this lesion caused by infection or tumor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vertebral impingement due to wrist ulnar pain, patients who have undergone ulnar shortening surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-04-26 (Estimated); Study Completion 2019-04-26 (Estimated)

PRIMARY OUTCOMES:
4-Item Pain intensity Measure | 5 seconds
  Each item is scored 0-10(0=no pain;10=pain as bad as can be)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan